CLINICAL TRIAL: NCT02623387
Title: A Prospective Randomized Controlled Trial of Ultrasound Guided Versus Standard Paravertebral Blockade in Breast Surgery
Brief Title: Ultrasound Guided Versus Standard Paravertebral Blockade in Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, Deirdre Nally, Senior Registrar in General Surgery, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UHG15
Record Dates: First submitted 2015-11-26; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Regional Anaesthesia; Mastectomy; Breast-Conserving Surgery
Keywords: paravertebral block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Paravertebral Block (Active Comparator): Patients receiving a conventional paravertebral block of dilute local anaesthetic (eg. 5ml of 0.5% bupivacaine or similar) administered using anatomical landmarks
  Interventions: Procedure: Ultrasound guided paravertebral block
- Ultrasound Guided Paravertebral Block (Active Comparator): Patients receiving paravertebral block of dilute local anaesthetic (eg. 5ml of 0.5% bupivacaine or similar) administered under ultrasound guidance
  Interventions: Procedure: Ultrasound guided paravertebral block

INTERVENTIONS:
Procedure: Ultrasound guided paravertebral block — Paravertebral blocks is a regional anaesthetic technique in which thoracic spinal nerves are inhibited for post operative analgesia in patients undergoing breast surgery. The site of injection can be determined using anatomical landmarks (standard) or using ultrasound guidance.
  Other Names: US paravertebral block

SUMMARY:
The aim of this study is to compare conventional and ultrasound guided paravertebral blocks to with respect to efficacy, patient satisfaction and complication rates.

DETAILED DESCRIPTION:
Adequate pain control is important in breast cancer surgery. In addition to benefits to patients, effective pain management strategies also facilitate day case surgery. Regional anaesthetic techniques, and paravertebral blocks in particular, are valuable in this sphere. The conventional method of administering this block is blind and depends on anatomical landmarks for placement. Performing the block under US guidance provides real time imaging while advancing the needle. This might allow for a more accurate placement and hence a more effective block which would enhance pain relief and minimise complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing resectional breast surgery
* Benign or malignant indications for surgery

Exclusion Criteria:

* Previous spinal surgery
* Severe coagulopathy
* Allergies to local anaesthesia
* Localised infection at site of injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Analgesia requirements in 24 hours post op. | 24hours
  Non opiate and opiate analgesia (morphine equivalent) intake at 24hours post op

SECONDARY OUTCOMES:
Pain Scores | 1, 2 and 24 hours post operatively and 1 week post operatively
  Measured on Visual Analogue Scale or Verbal Numerical Rating Scale at 1, 2 and 24 hours post operatively and 1 week
Patient satisfaction | Up to 2 weeks post operatively
  1. Satisfaction Questionnaire
  2. SF 36 Questionnaire
Complications | Up to 2 weeks post operatively
  Any complication of the procedure experienced

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Galway, Galway, Co. Galway, Ireland